CLINICAL TRIAL: NCT02806661
Title: Comparison of Vagus Nerve-preserving Robot-assisted Distal Gastrectomy (RADG) and Conventional Robot-assisted Distal Gastrectomy for Advanced Gastric Cancer (AGC)
Brief Title: Comparison of Vagus Nerve-preserving RADG and Conventional RADG for AGC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yingxue Hao (Other)
Responsible Party: Sponsor-Investigator, Yingxue Hao, Professor, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADG160416
Record Dates: First submitted 2016-04-16; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Cancer
Keywords: Robotic surgery; Vagus nerve preserving
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VPRDG for AGC (Experimental): Vagus nerve-preserving Robot-assisted distal subtotal gastrectomy (VPRDG) with D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Vagus nerve-preserving Robot-assisted Gastrectomy
- CRDG FOR AGC (Active Comparator): Conventional Robot-assisted distal subtotal gastrectomy (CRDG) with D2 lymphadenectomy without preserving vagus nerve will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Conventional Robot-assisted Gastrectomy

INTERVENTIONS:
Procedure: Vagus nerve-preserving Robot-assisted Gastrectomy
  Arms: VPRDG for AGC
Procedure: Conventional Robot-assisted Gastrectomy
  Arms: CRDG FOR AGC

SUMMARY:
Through comparative observation of robot vagus nerve preserving distal gastric cancer radical surgery and conventional robot distal gastric cancer radical surgery (not reserved vagus nerve) operative and postoperative indicators, and evaluating the feasibility and safety of vagus nerve preserving distal gastric cancer radical surgery in advanced gastric cancer. Which can provide the evidences for the clinical development of the preserving function gastric cancer surgery.

DETAILED DESCRIPTION:
Compare the robot vagus nerve preserving distal gastric cancer radical surgery and conventional robot distal gastric cancer radical surgery (not reserved vagus nerve). Observe the operative and postoperative indicators, and evaluate the feasibility and safety of vagus nerve preserving distal gastric cancer radical surgery in advanced gastric cancer. Which can provide the evidences for the clinical development of the preserving function gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged less than 70 years and more than 18 years;
2. Underwent gastroscopy and biopsy - preoperative definite for advanced gastric cancer invasion depth is T2, T3;
3. The lesion is in the middle and lower stomach;
4. Magix routine upper gastrointestinal barium meal, endoscopic ultrasonography, abdominal CT and chest X ray examination, clearly no nerve invasion and adjacent organ invasion and distant metastasis;
5. The preoperative examination of lung, liver, heart, renal insufficiency, surgical contraindication;
6. The preoperative abdominal CT or abdominal ultrasound without biliary disease and gallbladder stones;
7. No history of gastrointestinal dysfunction and other malignant tumor history;
8. The patients voluntarily participate in the study and signed informed consent.

Exclusion Criteria:

1. Older than 70 years old or because of chemotherapy surgery and complications after intolerance;
2. The vagus nerve invasion or invasion of adjacent organs or confirmed the presence of distant metastasis;
3. Have a history of abdominal surgery or chemotherapy before surgery;
4. The recent cardiovascular hemorrhagic or ischemic disease;
5. The amount of abnormal glucose tolerance or diabetes;
6. Not suitable for robotic surgery, such as body short that mechanical arm can not have enough activity range;
7. The history of biliary calculi or gastrointestinal dysfunction;
8. The other is not suitable for receiving robot surgery;
9. Participated in other clinical studies in the last month;
10. Other researchers not suitable for participation in the study of (HIV infection and intravenous drug addict), or other effects of this clinical study results analysis of the situation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | up to 36 months
  Recurrence rate in 3 years after operating.

SECONDARY OUTCOMES:
3-years survival rate | up to 36 months
  Survival rate in 3 years after operating.
The rate of Calculus of gallbladder | up to 12 months
  The rate of gallbladder calculus in 1 year after operating, which is diagnosed by ultrasound.
Number of retrieving lymph nodes | up to 1 week
  The number of dissecting lymph nodes during operating.
Inflammatory factors | 6 h, 12 h, 24 h, and 72h after operating
  Detecting Interleukin -10 (IL-10), C-reactive protein (CRP) and Tumor Necrosis Factor (TNF-a) in 6 h, 12 h, 24 h, and 72h after operating.

CONTACTS AND LOCATIONS:
Overall Officials: Yingxue Hao, M.D., Principal Investigator — Southwest Hospital, Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Yes, the investigators can share the data with other.